CLINICAL TRIAL: NCT05704309
Title: Alzheimer's Disease and Alzheimer's Disease Related Dementias in Prediabetes and Type 2 Diabetes: The Diabetes Prevention Program Outcomes Study AD/ADRD Project
Brief Title: The Diabetes Prevention Program Outcomes Study AD/ADRD Project
Acronym: DPPOS-4
Status: Enrolling by invitation | Type: Observational
Sponsor: Marinella Temprosa (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor-Investigator, Marinella Temprosa, Principal Investigator, George Washington University
Organization: George Washington University (Other)
Other Study IDs: DPPOS AD/ADRD; 1U19AG078558 (NIH)
Record Dates: First submitted 2023-01-11; First posted 2023-01-30 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Diabetes; Alzheimer Disease; Dementia, Vascular; Dementia; PreDiabetes
MeSH Terms: conditions — Diabetes Mellitus; Alzheimer Disease; Dementia, Vascular; Dementia; Prediabetic State

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biospecimens for urine, plasma and serum stored and banked from 2 visits
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The DPPOS AD/ADRD project will address the overarching question: What are the determinants and the nature of cognitive impairment among persons with pre-diabetes (PreD) and type 2 diabetes (T2D), who are a high-risk group for cognitive impairment and represent a large fraction of the United States (US) population? This U19 proposal addresses the National Alzheimer's Project Act goal to "prevent, halt, or reverse AD" in the high-risk group of persons with pre-diabetes and type 2 diabetes, who represent over half of the population aged 60 years and older in the US.

DETAILED DESCRIPTION:
DPPOS AD/ADRD focuses on one of the most important, complex questions in Alzheimer's disease (AD) and Alzheimer's disease-related dementias (ADRD) research: What are the determinants and the nature of cognitive impairment among persons with pre-diabetes (PreD) and type 2 diabetes (T2D), who are a high-risk group for cognitive impairment and represent a large fraction of the United States (US) population? Despite knowledge that persons with PreD and T2D are a high-risk group for cognitive decline, mild cognitive impairment (MCI), and dementia, the risk factors, mechanisms, and neuropathology of cognitive impairment in persons with PreD and T2D remain unclear. Gaps in knowledge on cognitive impairment in PreD and T2D include: (a) the role of AD and/or non-AD neuropathology beyond vascular contributions to cognitive impairment and dementia (VCID); (b) the role of glycemia, related metabolic factors such as hyperinsulinemia, and traditional micro and macrovascular complications of PreD/T2D; (c) the role of glucose-lowering medications, primarily metformin; and (d) the role of physical activity, physical function, and frailty, key in PreD and T2D. The 4 interrelated projects will address these gaps, leveraging the Diabetes Prevention Program (DPP) Outcomes Study (DPPOS) cohort and its detailed PreD/T2D phenotyping, adding state of the art AD/ADRD phenotyping. The DPPOS cohort currently has a mean age of 72 years, with 76% over the age of 65. Thus, the cohort is in a period of the lifespan when the development of cognitive decline, MCI, and dementia accelerates. This extensively phenotyped cohort represents an estimated 50 million Americans. To address this proposal's complex interrelated questions, the study has two waves of state-of-the-art AD/ADRD phenotyping during the proposed 5-year funding period, including comprehensive cognitive assessments and syndrome adjudication and plasma and brain imaging biomarkers of AD/ADRD. The study will address the complex overarching question of our project through the following aims: (1) To establish 5 cores to support the 4 integrated scientific projects: An Administrative Core, a Clinical Operations and Procedures Core, a Cognitive Assessment and Adjudication Core, a Neuroimaging and Plasma Biomarkers Core, and A Biostatistics and Data Infrastructure Core: (2) To conduct 4 integrated projects focused on key aspects of the central question of this proposal: Project 1 will examine the association of cognitive decline, MCI, and dementia in the DPPOS cohort with biomarkers of neuropathology and brain insulin signaling, and with sociodemographic and behavioral factors; Project 2 will examine the associations of cumulative glycemia, related metabolic factors, and microvascular and macrovascular complications, with cognitive syndromes and biomarkers of neuropathology; Project 3 will examine the association of cumulative exposure to metformin and other T2D medications with cognitive syndromes and biomarkers of neuropathology; Project 4 will evaluate the association of trajectories of physical activity, physical function and frailty with cognitive syndromes and biomarkers of neuropathology.

ELIGIBILITY:
Inclusion Criteria:

* All surviving participants originally randomized in the Diabetes Prevention Program
* For Brain Imaging subcohort, only participants aged 55 years and older and those without contraindication to MRI will be included. Contraindications to MRI include the inability to lie flat, claustrophobia, and the presence of indwelling metallic objects, medical or non-medical, that are not 3T MRI compatible.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The DPPOS (2002-2022) is a 25-center observational study that started as the DPP randomized controlled clinical trial (1996-2001). The DPP demonstrated the ability to reduce the development of T2D with intensive lifestyle or metformin compared with placebo among persons with PreD. The combined DPP and DPPOS have followed the original DPP cohort for a mean of 23 (range 21-25) years as of 2022. For this project, we expect that the cohort will have 1979 participants, with approximately two thirds with T2D of precisely known duration. Forty-eight percent of the cohort are ethnic and racial minorities that are at relatively higher risk of AD/ADRD compared with non-Hispanic whites, and 71% are women.
Sampling Method: Non-Probability Sample
Enrollment: 1976 (Estimated)
Dates: Start 2022-11-07 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Cognitive Diagnoses | Sept 2022 to October 2026
  Classification of normal, mild cognitive impairment or dementia based on NACC UDS

SECONDARY OUTCOMES:
ptau-181 | Sept 2022 to October 2026
  Plasma biomarkers for AD/ADRD
Aβ42/40 ratio | Sept 2022 to October 2026
  Plasma biomarkers for AD/ADRD
Neurofilament Light Chain (NfL) | Sept 2022 to October 2026
  Plasma biomarkers for AD/ADRD
Glial fibrillary acidic protein (GFAP) | Sept 2022 to October 2026
  Plasma biomarkers for AD/ADRD
Amnestic cognitive decline | Sept 2022 to October 2026
  Based on the SEVLT immediate recall (sum of trials 1-3) and delayed recall (trial 4)
Non-amnestic cognitive decline | Sept 2022 to October 2026
  DSST measure
White matter microstructure | March 2023 to October 2026
  Among ppts in the neuromaging subcohort

CONTACTS AND LOCATIONS:
Overall Officials: Jose Luchsinger, Principal Investigator — Columbia University; David Nathan, Study Chair — Massachusetts General Hospital; Marinell Temprosa, Principal Investigator — George Washington University
Locations (27):
- United States (27):
  - SW American Indian Center - Phoenix, Phoenix, Arizona
  - University of California Los Angeles, Alhambra, California
  - University of California San Diego, San Diego, California
  - University of Colorado, Aurora, Colorado
  - Medstar Health Research Institute, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - University of Hawaii, Honolulu, Hawaii
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Pennington Biomedical Center, Baton Rouge, Louisiana
  - Johns Hopkins University, Lutherville, Maryland
  - Biostatistics Center, George Washington University, Rockville, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Joslin Diabetes Center, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - University of New Mexico, Albuquerque, New Mexico
  - SW American Indian Center - Shiprock, Shiprock, New Mexico
  - SW American Indian Center - Zuni, Zuni, New Mexico
  - Columbia University Medical Center, New York, New York
  - Columbia University, New York, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Tennessee, Memphis, Tennessee
  - University of Texas Health Science Center San Antonio, San Antonio, Texas
  - University of Washington, VA Puget Sound Health Care System, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
We will have data in the NACC (National Alzheimer's Coordinating Center) data repository for NACC UDS (Uniform Data Set) data and the rest will be available in the NIDDK data repostiory
Supporting Information: Study Protocol
Time Frame: NACC 2025 and 2027 NIDDK repository 2027
Access Criteria: Available to public by application
URL: https://dppos.bsc.gwu.edu/web/dppos/data

REFERENCES:
- See also: Study website — http://www.dppos.org
- Available data/document: Individual Participant Data Set: DPPOS — https://repository.niddk.nih.gov/studies/dppos/
- Available data/document: Individual Participant Data Set — https://naccdata.org/requesting-data/data-request-process — will be available in 2025